CLINICAL TRIAL: NCT04243005
Title: Supramarginal Resection in Patients With Glioblastoma: A Randomised Controlled Trial
Brief Title: Supramarginal Resection in Glioblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Odense University Hospital (Other); Sahlgrenska University Hospital (Other); Turku University Hospital (Other Government); Karolinska University Hospital (Other); Norwegian University of Science and Technology (Other); Uppsala University Hospital (Other); University Hospital, Umeå (Other); Haukeland University Hospital (Other); Ullevaal University Hospital (Other); Rikshospitalet University Hospital (Other); Tampere University Hospital (Other); Helsinki University Central Hospital (Other); Kuopio University Hospital (Other); Oulu University Hospital (Other); Medical University of Vienna (Other); Paracelsus Medical University (Other); Medical Center Haaglanden, The Hague, The Netherlands (Unknown); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/1046
Record Dates: First submitted 2020-01-08; First posted 2020-01-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
Keywords: Neurosurgical procedures
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked until postoperative period. Outcome assessor will be masked until all predefined outcomes have been analysed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional surgery (Active Comparator): Aim of gross total resection (i.e. removal of contrast enhancing tumor) according to institutional practice. No limit in use of technical adjuncts in this arm.
  Interventions: Procedure: Conventional surgery
- Supramarginal surgery (Experimental): Aim of supramarginal resection, where a margin of at least 10 mm is considered feasible prior to surgery. The resection is guided by the T2 volume (i.e. zone of edema) where removal of as much as possible of this zone (or beyond) is attempted as long as considered safe
  Interventions: Procedure: Supramarginal resection

INTERVENTIONS:
Procedure: Supramarginal resection — Aim of supramarginal resection, where a margin of at least 10 mm is considered feasible prior to surgery. The resection is guided by the T2 volume (i.e. zone of edema) where removal of as much as possible of this zone (or beyond) is attempted as long as considered safe
  Arms: Supramarginal surgery
Procedure: Conventional surgery — Aim of gross total resection (i.e. removal of contrast enhancing tumor) according to institutional practice. No limit in use of technical adjuncts in this arm.
  Arms: Conventional surgery

SUMMARY:
Gliomas are the most common malignant brain tumor. Glioblastoma, WHO grade IV astrocytoma, is the most common subtype and unfortunately also the most aggressive subtype with median survival in population based cohorts being only 10 months. Extensive surgical resections followed by postoperative fractioned radiotherapy and concomitant and adjuvant temozolomide prolong survival and is the standard treatment.

The investigators think there is significant potential in individualized surgical decision-making in glioblastoma management. The idea that some patients are amendable to radical surgery, while others should be treated more conservatively, is not controversial in other fields of oncology. The current concept in all patients with glioblastoma is "maximum safe resection of the contrast enhancing tumor", but this may in selected cases be extended to simply "maximum safe resection" tailored to the patient and extent of disease at hand.

Densely proliferating tumor cells have been found from at an average of 10 mm beyond the margins of contrast enhancement in high-grade gliomas. There are now several case series, using various definitions of supramarginal resection, but they have in common that they report a benefit of resection with a margin. This potential benefit also comes together with an associated neurological risk, making this approach unethical and simply not feasible in the patients with glioblastoma as a whole.

Objective of this study is: To investigate if resection with a margin, that is significantly beyond the radiological contrast enhancement, improves survival in selected patients with glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. A suspected diagnosis of supratentorial glioblastoma by MRI.(A)
2. Indication for surgical treatment and where supramarginal resection is considered possible according to the preoperative imaging. This consideration needs to be verified by two specialists in neurosurgery.
3. Negative work-up for other primary tumor(B)
4. Karnofsky performance status of 70 - 100.

A) If randomized to supramarginal surgery, intraoperative frozen section must conclude with "high-grade glioma" to be able to proceed. Surgery in two sessions is also possible in supramarginal group if there is no intraoperative frozen section available or frozen section indicate another diagnosis, but final histopathology reveals a glioblastoma. In case of surgery in two session, there must be no more than 30 days between procedures. See flow-chart in attachment 1.

B) No suspected primary tumor seen on CT chest, abdomen and pelvis. If relevant symptoms/clinical suspicion also supplement with mammography, dermatologist exam, relevant endoscopies etc.

Exclusion Criteria:

1. Not willing to be randomized.
2. Informed consent not possible (e.g. language barriers, aphasia, cognitive severely impaired).
3. Contrast enhancement volume bilateral OR involving corpus callosum.
4. Contrast enhancement along the ependymal lining of ventricles (contact is however not an exclusion criteria).
5. Contrast enhancement involving several lobes.
6. History of major psychiatric disorder such as psychosis, schizophrenia and/or mood disorder (e.g. depression and bipolar disorder) in need of hospitalization
7. Unfit for participation for any other reason judged by the including physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 36 months after the last included patient.
  Overall survival according to intention-to-treat

SECONDARY OUTCOMES:
Proportion alive | 24 months after randomization.
  Proportion alive
Proportion alive | 36 months after randomization.
  Proportion alive
Neurological function | Early postoperative (i.e. prior to radiotherapy) to 36 months
  Neurological assessment in Neuro-Oncology (NANO) Scale is a tool used by healthcare providers to objectively quantify the impairment caused by a tumor within the central nervous system. The NANO is composed of 9 items. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NANO scale score. The maximum possible score is 23, with the minimum score being a 0.
Health-related quality of life assessed by EQ-5D 3L | Early postoperative (i.e. prior to radiotherapy) to 36 months
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Health-related quality of life assessed by EORTC QLQ C30 | Early postoperative (i.e. prior to radiotherapy) to 36 months
  The QLQ-C30 is a cancer health-related quality-of-life questionnaire that has been widely used in clinical trials and investigations using PROs for individual patient management. It includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality-of-life and financial impact. Subjects respond on a four-point scale from "not at all" to "very much" for most items. Most items use a "past week" recall period. Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of function and higher levels of symptom burden.
Health-related quality of life assessed by BN20 | Early postoperative (i.e. prior to radiotherapy) to 36 months
  The European Organization for Research and Treatment of Cancer (EORTC) QLQ-BN20 is a quality of life assessment specific to brain neoplasms. Consists of 20 items that assess future uncertainty, visual disorder, motor dysfunction, and communication deficit. Items are presented as questions on a scale ranging from 1 = "not at all" to 4 = "very much." Higher score means worse outcome.
Neurocognition | Early postoperative (i.e. prior to radiotherapy) to 36 months
  The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It examines functions including registration (repeating named prompts), attention and calculation, recall, language, ability to follow simple commands and orientation. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
Surgical complication | 30 days
  surgical complication grade 3, 4 and 5, assessed using the Dindo-Clavien classification
Proportion with contrast remnant | Within 72 hours postoperative
  Resection proportion with contrast remnant
Extent of resection, T2/FLAIR remnant | Within 72 hours postoperative
  Proportion with remnant in terms of hyper intensity changes in T2/FLAIR
Margin of resection | Within 72 hours postoperative
  Cavity volume/contrast enhancement volume

OTHER OUTCOMES:
Overall Survival; as treated | 36 months after the last included patient.
  Accounting for cross-over or failure to achieve predefined surgical aim. "As treated" populations when no margins in supramarginal group and unintended contrast remnant in group aiming at conventional gross-total resection or even if significant supramarginal resection in this group

CONTACTS AND LOCATIONS:
Overall Officials: Asgeir S Jakola, MD, PhD, Principal Investigator — St.Olavs University Hospital and Sahlgrenska University Hospital; Geir Bråthen, MD, PhD, Study Director — St. Olavs Hospital
Locations (17):
- Medical University of Vienna, Vienna, Austria
- Odense University Hospital, Odense, Denmark
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - Haaglanden MC, The Hague
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Rikshospitalet, Oslo
  - Ullevål University Hospital, Oslo
  - St Olavs Hospital, Trondheim
- Sweden (4):
  - Sahlgrenska University Hospital,, Gothenburg
  - Karolinska University Hospital, Stockholm
  - University Hospital of Umeå, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No